CLINICAL TRIAL: NCT06507735
Title: The Effects of Mannose Supplementation on Glycosylation and Protein Levels in Human Sera
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey SoRelle, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU-2024-0127; Velos Study Number (Other: 58400)
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Physiological Stress
MeSH Terms: interventions — Mannose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mannose supplementation (Experimental): Mannose supplementation will be given and subjects will be studied at baseline and after treatment.
  Interventions: Dietary Supplement: Mannose

INTERVENTIONS:
Dietary Supplement: Mannose — Mannose is a sugar monomer that is important in the glycosylation of many proteins. The concentration of mannose in mammalian plasma is ~50-100 μM, which is primarily derived from N-glycan processing. Taking dietary mannose supplements can raise the levels of plasma mannose by 3- to 5-fold. There are currently no known adverse effects of mannose supplementation in humans.

SUMMARY:
The purpose of our study is to investigate the effects of supplemental mannose on sera of humans who are healthy. We will perform proteomics studies to elucidate changes to glycan structure and protein level changes. We hypothesize that we may find that mannose supplies more properly glycosylated protein substrate and helps expedite protein synthesis, that excess mannose leads to alternative glycan structures which confer improved stability, or that there are new sites that become glycosylated after mannose supplementation.

DETAILED DESCRIPTION:
Subjects will be enrolled and a baseline blood sample taken. Subjects will take mannose supplements for 1 week (3-4 packets of a standard dose in water), then a follow up blood sample will be taken.

Subject blood will be analyzed by proteomic analysis for 1) change in glycan structure or 2) other protein based approaches to measure changes in levels of proteins.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* No known medical conditions
* Taking no medications or nutritional supplements
* Agree to the study and provide informed consent

Exclusion Criteria:

* Less than 18 years of age
* Known medical diagnosis, including pregnancy
* Presently taking medications and/or nutritional supplements
* Do not provide consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Changes to glycan structure | ~1 month
  Glycopeptide mass spectrometry will be applied to the major glycoproteins present in serum.
Change in glycoprotein levels | ~1 month
  Standard laboratory methods such as ELISA in either research or clinical laboratory settings (Roche Cobas or similar platform).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey SoRelle, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No